CLINICAL TRIAL: NCT03178903
Title: tDCS for Increasing Exercise Adherence in Individuals With Elevated Depressive Symptoms
Brief Title: tDCS for Increasing Exercise Adherence in Depressed Individuals
Acronym: StRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1608-002; R21CA214102 (NIH)
Record Dates: First submitted 2017-05-10; First posted 2017-06-07 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-01

CONDITIONS: Depression; Physical Activity
MeSH Terms: conditions — Depression; Motor Activity | interventions — Transcranial Direct Current Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS and Aerobic Exercise (Active Comparator): Each participant will undergo a 20-minute session of transcranial direct current stimulation (tDCS) delivered to the dorsolateral prefrontal cortex (DLPFC). Each session of tDCS will be immediately followed by a supervised 30-minute, moderate-intensity bout of exercise. These procedures will occur 3x/week for 8 weeks.
  Interventions: Other: tDCS; Behavioral: Aerobic Exercise (AE)
- Sham tDCS and Aerobic Exercise (Sham Comparator): Each participant will undergo a 20-minute session of sham transcranial direct current stimulation (tDCS) delivered to the dorsolateral prefrontal cortex (DLPFC). Each session of tDCS will be immediately followed by a supervised 30-minute, moderate-intensity bout of exercise. These procedures will occur 3x/week for 8 weeks.
  Interventions: Other: Sham tDCS; Behavioral: Aerobic Exercise (AE)

INTERVENTIONS:
Other: tDCS — Participants in transcranial direct current stimulation (tDCS) will receive tDCS over the dorsal-lateral prefrontal cortex for 20 minutes, 3 times per week for 8 weeks.
  Arms: tDCS and Aerobic Exercise
Other: Sham tDCS — Participants in sham transcranial direct current stimulation (tDCS) will receive shame tDCS over the dorsal-lateral prefrontal cortex for 20 minutes, 3 times per week for 8 weeks.
  Arms: Sham tDCS and Aerobic Exercise
Behavioral: Aerobic Exercise (AE) — Participants will engage in supervised, 30-minute bouts of moderate-intensity exercise 3x/week for 8 weeks.

SUMMARY:
The purpose of this study is to examine the efficacy of tDCS (transcranial direct current stimulation) for increasing exercise adherence among low active individuals with elevated depressive symptoms. The investigators expect that this project will contribute much needed knowledge about the role that tDCS can play in changing the affective experience of exercise.

DETAILED DESCRIPTION:
Exercise adherence is a significant public health problem. Affective experiences during exercise predict long-term physical activity (PA) levels. Therefore, approaches to improving the affective experience of exercise are both important and likely to have high impact. This may be particularly true among individuals with elevated depressive symptoms due to their tendency toward more negative and less positive affect. tDCS is a noninvasive brain stimulation approach with a growing body of literature supporting its effects on cognitive and emotional processing in varied populations, including some support for those with depression. In addition, there is recent increased interest in utilizing tDCS in the context of exercise (see above) and in obesity prevention. While the effects of tDCS on behavioral and cognitive functioning are still developing, promising findings have emerged for tDCS used in repeated combination with a behavioral or cognitive intervention. Given that tDCS is relatively safe, inexpensive, and portable, individuals who struggle with enjoying exercise could be afforded a practical option for increasing and maintaining physical activity levels.

We propose to conduct a pilot randomized controlled trial of tDCS versus sham delivered 3x/week for 8 weeks in the context of a supervised aerobic exercise (AE) program among 72 low-active individuals with elevated depressive symptoms. Follow-up assessments will be conducted at end of treatment, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 65 years of age
* be low active
* have elevated levels of depressive symptoms
* interested in starting an exercise program in the next month

Exclusion Criteria:

* history of mania or hypomania
* current psychotic disorder
* current DSM-5 diagnosis of an eating disorder
* DSM-5 moderate and severe substance use disorder
* current suicidality or homicidality
* current DSM-5 diagnosis of major depressive disorder that is not currently being treated with pharmacotherapy or psychotherapy
* physical disabilities or medical problems that would prevent participation in moderate intensity exercise or may be contraindicated for tDCS
* current pregnancy or intent to become pregnant during the next 8 weeks
* pacemaker or metal implanted in the cranial cavity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS and Aerobic Exercise | Sham tDCS and Aerobic Exercise
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS and Aerobic Exercise | Sham tDCS and Aerobic Exercise | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9.7) | 50.1 (11.1) | 49.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 23 | 46
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Baseline depressive symptoms were collected using the Center for Epidemiological Studies--Depression (CES-D) measure. The range of scores is 0 to 60. Scores above 15 indicate clinical depression. Higher scores indicate higher levels of depression.
  units on a scale | 22.9 (10.0) | 21.8 (11.6) | 22.3 (10.7)
Minutes of Moderate-to-Vigorous Physical Activity (MVPA) [Mean (Standard Deviation); unit: minutes per day] | 14.9 (11.0) | 20.0 (14.4) | 17.4 (13.0)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Levels
Description: Accelerometry-based moderate-to-vigorous physical activity (MVPA)
Time Frame: 8 week assessment
Population: The numbers analyzed include only individuals that provided valid wear-time data on the primary outcome measure, using accelerometry. Specifically, only participants that provided 3 days of 8 hours/day valid wear time were included in the analysis of the primary outcome.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | tDCS and Aerobic Exercise | Sham tDCS and Aerobic Exercise
Number analyzed (Participants) | 19 | 17
minutes per day | 17.4 (9.8) | 21.0 (17.4)
Statistical Analysis 1: Comparison: tDCS and Aerobic Exercise vs Sham tDCS and Aerobic Exercise; Test type: Superiority; p = .87, ANCOVA — p<.05 was the a priori threshold for statistical significance; Covarying for baseline depressive symptoms and MVPA; Mean Difference (Final Values) = .678

ADVERSE EVENTS:
Time Frame: 6 months
Description: It does not differ from clinicaltrials.gov definitions
Arm/Group | tDCS and Aerobic Exercise | Sham tDCS and Aerobic Exercise
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 4/25 | 0/26
Other Adverse Events (participants affected / at risk) | 2/25 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS and Aerobic Exercise (N=25) | Sham tDCS and Aerobic Exercise (N=26)
Psychiatric Inpatient Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
Medical Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical Hospitalization (Cardiac disorders) | 1 (1) | 0 (0)
Medical Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS and Aerobic Exercise (N=25) | Sham tDCS and Aerobic Exercise (N=26)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
knee injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT03178903/Prot_SAP_ICF_000.pdf